CLINICAL TRIAL: NCT07252518
Title: Effect of Pentoxifylline Plus Coenzyme Q10 Combination Therapy Compared to Coenzyme Q10 Alone on Sperm Motility in Sub-fertile Male With Asthenozoospermia
Brief Title: Effect of Pentoxifylline + CoQ10 vs CoQ10 Alone on Sperm Motility in Subfertile Men With Asthenozoospermia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mst.Sumyara Khatun (Other)
Collaborators: Bangladesh Medical University (Other)
Responsible Party: Sponsor-Investigator, Mst.Sumyara Khatun, Medical officer, Bangladesh Medical University
Organization: Bangladesh Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 5721
Record Dates: First submitted 2025-09-17; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-09

CONDITIONS: Asthenozoospermia
Keywords: Asthenozoospermia; Pentoxifylline; Coenzyme Q10
MeSH Terms: conditions — Asthenozoospermia | interventions — coenzyme Q10; Pentoxifylline; Tablets

STUDY DESIGN:
Intervention Model Description: Open label parralel design randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (PTX+ CoQ10) (Experimental): Participants receive pentoxifylline 400mg orally twice daily plus Coenzyme Q10 100mg twice daily orally
  Interventions: Combination Product: Pentoxifylline 400 MG Oral Tablet
- Active Comparator (Coenzyme Q10) (Active Comparator): Participants receive Coenzyme Q10 100mg twice daily orally
  Interventions: Dietary Supplement: Coenzyme Q 10

INTERVENTIONS:
Dietary Supplement: Coenzyme Q 10 — Participants will receive Coenzyme Q10 100 mg twice daily for 3 months
  Arms: Active Comparator (Coenzyme Q10)
Combination Product: Pentoxifylline 400 MG Oral Tablet — Participants will receive pentoxifylline 400mg twice daily plus coenzyme Q10 100mg twice daily for 3 months
  Other Names: Coenzyme Q10
  Arms: Experimental (PTX+ CoQ10)

SUMMARY:
The goal of this clinical trial is to learn if drug Pentoxifylline plus Coenzyme Q10 work to treat asthenozoospermia in subfertile male. It will also learn about the safety of drug Pentoxifylline plus Coenzyme Q10. The main questions it aims to answer are:

Does drug Pentoxifylline plus Coenzyme Q10 increase the motility of sperm in participants? What medical problems do participants have when taking drug Pentoxifylline plus Coenzyme Q10 ? Researchers will compare drug Pentoxifylline plus Coenzyme Q10 combination to Coenzyme Q10 alone to see if drug Pentoxifylline plus Coenzyme Q10 combination works better.

Participants will:

Experimental Group:Pentoxifylline 400mg twice dailyand Coenzyme Q10 100mg twice daily for 3 months.

Comparator Group: Coenzyme Q10 100mg twice daily for 3 months Visit the clinic after three months of treatment for checkups and tests

DETAILED DESCRIPTION:
This Randomized controlled trial will be conducted in the Department of Reproductive Endocrinology & Infertility, BMU from the day of approval. Ethical clearance will be obtained from the Institutional Review Board. A total 56 sub-fertile men with asthenozoospermia (Total motility 20% to <42%), according to WHO Laboratory manual 6th Edition in 2021, fulfilling the inclusion and exclusion criteria.will be approached for informed written consent after discussing the purpose and procedure of the study. Participants will be recruited from our OPD-2, room no-301 and referred outdoor room no-108, department of Reproductive Endocrinology & Infertility.Baseline infertility investigations and semen analysis will be done. Detailed socio-demographic data, history, and investigations will be recorded in a predesigned data sheet. Eligible men who will give their informed consent will be randomized to either. Random sequence generation will be done by someone not involved in the study. Allocation concealment will be done by serially numbered closed opaque envelopes. Each envelope will be labeled with a serial number and will have a card noting the intervention type. Allocation will never be changed after opening the closed envelopes.At baseline, a minimum of two specimen will be collected at 4 weeks intervaland the second results showing asthenozoospermia will be considered as the baseline results.Semen sample will be collected after maintaining 3-5 days of abstinence, in the semen collection room no-110 of Reproductive Endocrinology & Infertility, BMU by masturbation in a sterile plastic container. After getting the samples, they will be allowed to liquefy at 37 degrees Celsius and then will be analyzed according WHO,2021, in the laboratory of Reproductive Endocrinology & Infertility department. The sperm parameter will be checked by Makler Counting Chamber. An aliquot (0.5 ml) of each well-mixed semen sample will be placed on the Makler counting chamber, and the coverslip will be applied. Motility evaluation will be performed within 3-5 minutes after application of the sample to avoid errors due to tendency of sperm to migrate from the periphery. All non-motile sperms will be counted within 9 or 16 squares. Then motile sperms will be counted in the same area and the grade of motility will be estimated from +1 to +4. This procedure will be repeated in another area of the grid,as well as from another 3-4 drops and the average will be calculated.

Experimental Group will receive (Pentoxifylline 400mg and Coenzyme Q10 100mg) twice daily and ComparatorGroup will receive (Coenzyme Q10 100mg) twice daily for 3 months. They will be informed not to take other medications that could affect spermatogenesis during the study period expect after counseling physician.

ELIGIBILITY:
Inclusion Criteria:

* Sub fertile men with asthenozoospermia(Total motility20% to less than 42%) according to WHO semen analysis,2021.
* Age 20-50 years.

Exclusion Criteria:

* Severe oligoasthenoteratozoospermia
* Any medical, endocrine and genetic disorders, history of chemotherapy or radiotherapy, genital infection, genital surgery.
* Antioxidants supplmentation in the last 3 months
* Drug, alcohol or substance abuse, psycho-sexual abnormalities.
* Any known hypersensitivity to xanthine related product, recent cerebral or retinal haemorrhage Severe oligoasthenoteratozoospermia
* Any medical, endocrine and genetic disorders, history of chemotherapy or radiotherapy, genital infection, genital surgery.
* Antioxidants supplmentation in the last 3 months
* Drug, alcohol or substance abuse, psycho-sexual abnormalities.
* Any known hypersensitivity to xanthine related product, recent cerebral or retinal haemorrhage

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 56 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Progressive sperm motility | Baseline(pre treatment) and 12 weeks after start
  Percentage of sperm showing progressive motility (WHO catagories A+B) on microscopic examination,measured using WHO manual standards,after 30-60 minutes liquefaction, at 37 degree celcius, averaged over two independent readings by trained laboratory technicians blinded to treatment allocatiob

SECONDARY OUTCOMES:
Total sperm motility | Baseline (pre treatment) and 12 weeks after start of treatment
  Percentage of motile sperm (WHO catagories A+B+C) measured on fresh semen samples using WHO semen analysis method (latest edition) .Total motility is the percentage of sperm showing any motility (progressive and non progressive ) at the time of analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Jesmine Banu, MS, Principal Investigator — Bangladesh Medical University
Locations (1):
- Bangladesh Medical University, Dhaka, Shahbag, Bangladesh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alahmar AT. The effects of oral antioxidants on the semen of men with idiopathic oligoasthenoteratozoospermia. Clin Exp Reprod Med. 2018 Jun;45(2):57-66. doi: 10.5653/cerm.2018.45.2.57. Epub 2018 Jun 29. PMID 29984205
- [Background] Barbonetti A, Tienforti D, Castellini C, Giulio FD, Muselli M, Pizzocaro A, Vena W, Baroni MG, Pivonello R, Isidori AM, Maggi M, Corona G. Effect of antioxidants on semen parameters in men with oligo-astheno-teratozoospermia: a network meta-analysis. Andrology. 2024 Mar;12(3):538-552. doi: 10.1111/andr.13498. Epub 2023 Jul 26. PMID 37495550